CLINICAL TRIAL: NCT07217769
Title: Effects of Operational Naps on Blood Pressure and Performance Among Night Shift Workers
Acronym: EONN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Daniel Patterson, PhD, NRP, Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY25070009; R61HL172984 (NIH)
Record Dates: First submitted 2025-10-02; First posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Shift Work
Keywords: Night shift; Sleep; Napping; Blood pressure; Psychomotor performance; Sleep inertia; Caffeine
MeSH Terms: conditions — Idiopathic Hypersomnia

STUDY DESIGN:
Intervention Model Description: This study uses an incomplete block design with participants completing 4 of the 5 conditions in random order.
Masking Description: Participants are blinded to the nap duration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Napping order (Other): 5 x 4 x 3 x 2 = 120 possible orderings of the 5 interventions for each person.
  Interventions: Behavioral: No-nap; Behavioral: 15-min nap; Behavioral: 30-min nap; Behavioral: 45-min nap; Behavioral: 60-min nap

INTERVENTIONS:
Behavioral: No-nap — No-nap opportunity offered
Behavioral: 15-min nap — A 15-minute nap opportunity at 02:00am
Behavioral: 30-min nap — A 30-minute nap opportunity at 02:00am
Behavioral: 45-min nap — A 45-minute nap opportunity at 02:00am
Behavioral: 60-min nap — A 60-minute nap opportunity at 02:00am

SUMMARY:
Night shift work schedules disrupt sleep and have a negative impact on cardiovascular health. Most who work in public safety occupations and in healthcare work night shifts. These workers experience abnormal blood pressure during night shifts and are at greater risk of cardiovascular disease. Napping during night shifts can help to restore blood pressure patterns to a more normal pattern and may help to reduce risk of cardiovascular disease. Naps may also have an impact on alertness and performance immediately upon waking. The overarching goal of this study is to determine which duration of a nap taken during simulated night shift work has the greatest impact blood pressure and post-nap performance.

Researchers will compare 5 nap durations to see which has the greatest impact on blood pressure patterns and post-nap psychomotor performance.

Researchers hypothesize that longer naps will lead to improved blood pressure outcomes and shorter naps will contribute to better performance after waking.

Findings will help employers and employees who work night shifts determine how best to incorporate brief naps during night shift work.

DETAILED DESCRIPTION:
Blunted blood pressure (BP) dipping is a well-described risk factor for cardiovascular disease (CVD) among older adults and individuals with chronic disease. Previous research shows that night shift workers are at risk and repeatedly exposed to blunted BP dipping as a consequence of sleep loss and irregular sleep. While occasional episodes of blunted BP dipping may not be harmful, repetitive exposure over years of night shift work, as experienced by public safety workers (PSWs) and healthcare workers (HCWs), is likely detrimental to cardiovascular health and increases risk of CVD. Recent research shows that exposure can be mitigated with brief on-duty naps, which briefly restore normal BP dipping. Despite these data, there is legitimate clinical equipoise regarding the optimal on-duty nap duration (dose) needed to maximize BP dipping and minimize threats to post-nap psychomotor performance (i.e., sleep inertia).

This study will use a Phase II, within subject, crossover, incomplete block randomized trial design to test the efficacy of 5 overnight on-duty nap conditions: no-nap, 15, 30, 45, and 60-minutes. The primary outcome is the proportion of participants with a clinically meaningful greater than or equal to 10% dip in BP during nap opportunities. The secondary outcome is focused on deficits in psychomotor performance at greater than or equal to 10 mins post-nap: a safety-critical moment for PSWs and HCWs.

Goal enrollment is set at 130, accounting for attrition. Each condition begins with 36 hours of at-home monitoring with non-invasive devices. The last 12 hours of each condition includes a 12-hour simulated night shift with nap opportunities provided at 0200 hours with the nap duration determined by the randomization schema. During the simulated night shift, participants will be continuously monitored with non-invasive devices, allowed to consume controlled amounts of caffeine, and complete standardized tests of psychomotor performance. Participants will be blinded to nap duration and caffeine dose. Volunteer participants will be asked to complete 4 of the 5 nap conditions.

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant adults (>18 years of age)
* certified public safety/healthcare shift worker
* is an active shift worker
* resides within the Western Pennsylvania region within reasonable driving distance

Exclusion Criteria:

* current use of medication for cardiovascular disease (e.g., hypertension)
* prior or current diagnosis of sleep apnea, narcolepsy, restless leg syndrome, ischemic heart disease, heart failure, stroke, chronic kidney disease, chronic liver disease, rheumatologic disease requiring prescription medication, and cancer requiring treatment in past 2 years
* undiagnosed severe sleep apnea (Apnea-Hypopnea Index >30) based on at-home test
* Abstains from caffeine or reports adverse effects from caffeine use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2030-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
BP dipping | During simulated night shift, 12 hours
  The ratio of mean sleep to mean wake blood pressure (BP) by taking the difference between the mean systolic blood pressure (SBP) and diastolic blood pressure (DBP) during nap opportunities, and the mean SBP and DBP during wake periods.
Psychomotor performance post-nap | During simulated night shift, greater than or equal to 10 minutes post intervention nap
  Severe psychomotor impairment post-nap as measured by the Psychomotor Vigilance Test Brief (PVT-B)

SECONDARY OUTCOMES:
Performance on simulated patient scenarios | During simulated night shift, 12 hours
  Change in performance pre-to-post nap. Performance rated from 0-100 with higher scores indicating better performance. Positive change indicates improved performance.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Patterson, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: No later than 3 years after completing the last follow-up of the last participant.
Access Criteria: Access through NHLBI BioLINCC repository